CLINICAL TRIAL: NCT00952432
Title: A Single-center, Prospective, Randomized, Positive Controlled, Parallel Design Trial to Compare the Efficacy of Acupuncture Therapy and Carbamazepine Oral Dosage in Patients With Carpal Tunnel Syndrome by Multiple Excitability Test
Brief Title: Compare the Efficacy of Acupuncture Therapy and Carbamazepine Oral Dosage in Patients With Carpal Tunnel Syndrome by Multiple Excitability Test
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Taipei Medical University WanFang Hospital (Other)
Responsible Party: Jia-Ying Sung, Wan Fang Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2008WFCRC-07
Record Dates: First submitted 2009-08-03; First posted 2009-08-06 (Estimated); Last update posted 2011-04-12 (Estimated); Status verified 2011-04

CONDITIONS: Carpal Tunnel Syndrome; Multiple Excitability Test
Keywords: Carpal Tunnel Syndrome; Multiple Excitability Test; Nerve Conduction Study; QtracW; carbamazepine; Acupuncture
MeSH Terms: conditions — Carpal Tunnel Syndrome | interventions — Carbamazepine; Acupuncture Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- ACUPUNCTURE (Active Comparator): ACUPUNCTURE
  Interventions: Procedure: Acupuncture
- MEDICATION (Active Comparator): Carbamazepine
  Interventions: Drug: Carbamazepine

INTERVENTIONS:
Drug: Carbamazepine — Carbamazepine 200mg, 1/2 tablet, TID for 1 month
  Arms: MEDICATION
Procedure: Acupuncture — Acupuncture
  Arms: ACUPUNCTURE

SUMMARY:
The goal of the study is to utilize BCTQ(Boston Carpal Tunnel Questionnaire), VAS (Visual Analog Scale), NCS (Nerve Conduction Study), and MET(Multiple Excitability Test) to evaluate and compare the efficacy of Acupuncture Therapy and Carbamazepine in Patients with Carpal Tunnel Syndrome.

ELIGIBILITY:
Inclusion Criteria:

* Age greater than 20 years old
* outpatient or inpatient subject with numbness of arm, clinically met diagnostic criteria of AAEM(American association of Electrodiagnostic Medicine CTS task force), and proven to have distal motor neurological disorder through nerve Conduction Study (distal motor latency >4.6 msec, decreased SNAP < 12uV or prolonged median sensory distal latency (palm to wrist) > 2.5msec)。
* Willing to sign the Informed Consent form

Exclusion Criteria:

* subject with external hand injury or disformation
* subject with Polyneuritis or Cervical nerve root lesions
* Subject with peripheral hypertrophy, hypothyroidism, multiple myeloma, or amyloidosis
* Allergic to Carbamazepine or similar type of medicine
* inability to act independently, or in the opinion of the investigator, not suitable for the study
* In the opinion of the investigator, the subject requires surgical repair of the Carpal Tunnel Syndrome, or the symptoms will be worsen result in irreversible damage to the subject if not treated with surgical repair within 3 months.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2009-05; Primary Completion 2011-05 (Estimated); Study Completion 2011-05 (Estimated)

PRIMARY OUTCOMES:
Use QtracW and NCS to evaluate the changes between pre-treatment and post-treatment in patients in both arms. | 12 weeks

SECONDARY OUTCOMES:
use BCTQ to evaluate the efficacy of 2 arms at week 4 and at week 12. | 12 weeks
use VAS to evaluate the efficacy of 2 arms at week 5, 8 and 12. | 12 weeks
Use Quality of Life questionnaire to compare the efficacy of 2 arms at week 12. | 12 weeks
Evaluate the safety of 2 arms during the study period | 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Jia-Ying Sung, MD, Principal Investigator — Taipei Medical University-Wan Fang Hospital
Locations (1):
- Taipei Medical University - Wan Fang Hospital, Taipei, Taiwan, Taiwan